CLINICAL TRIAL: NCT00000947
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Prophylaxis for Disseminated Mycobacterium Avium Complex Disease and Bacterial Pneumonia Versus Deferred Prophylaxis in HIV-Infected Patients Who Experience Rebound in CD4+ Cell Count Due to Active Antiretroviral Therapy
Brief Title: A Study to Evaluate the Effects of Azithromycin on MAC Disease Prevention in HIV-Positive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: CPCRA 048; 11600 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Placebos; Mycobacterium avium-intracellulare Infection; Acquired Immunodeficiency Syndrome; Antitubercular Agents; Azithromycin; Drug Resistance, Microbial; CD4 Lymphocyte Count; Antibiotics; Time Factors; Anti-HIV Agents; Pneumonia, Bacterial; Streptococcus pneumoniae
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; Pneumonia, Bacterial | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
This study is designed to find out whether HIV-positive patients whose immune systems have improved after receiving anti-HIV treatment should take azithromycin to prevent Mycobacterium avium complex (MAC) disease. This study also examines the possibility of putting off MAC prevention treatment in patients who respond well to anti-HIV drug therapy.

Azithromycin is approved for the prevention of MAC disease in people with HIV and low CD4 cell counts. However, some people who have taken azithromycin have been found to carry antibiotic-resistant bacteria (germs that can grow despite the presence of drugs used to kill them). It is not known whether the risks associated with taking azithromycin outweigh the risk of getting MAC disease.

DETAILED DESCRIPTION:
The need for MAC prophylaxis in advanced HIV disease is recognized. Prophylactic therapy is complicated, however, due to drug toxicity, potential drug interactions, patient noncompliance with multiagent regimens, microbial drug resistance, and high treatment costs. This study assesses the feasibility of deferring MAC prophylaxis in patients whose CD4+ cell counts rebound in response to antiretroviral therapy.

In this double-blind, placebo-controlled trial, patients are randomized to receive azithromycin weekly or matching placebo. Patients are switched to open-label azithromycin if they have an average CD4+ cell count less than 50 cells/mm3 on 2 consecutive counts obtained at least 48 hours apart (preferably no more than 60 days).

[AS PER AMENDMENT 10/23/97: SUBSTUDY CPCRA 054: A subset of participants of CPCRA 048 have oropharyngeal swabs taken at baseline and 4 months after randomization. Antibiotic susceptibility tests are then performed on isolates of S. pneumoniae.] [AS PER AMENDMENT 9/3/99: Participants in protocol version 3.0 are followed for data collection purposes every 4 months for 18 months until January 31, 2001. Data collection includes CD4 cell counts, viral RNA measurements, macrolide susceptibility in MAC isolates, and antibiotic susceptibility of isolates from bacterial pneumonia episodes.]

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have 2 CD4 counts over 100 cells/mm3 at least 30 days apart.
* Have a history of CD4 counts under 50 cells/mm3.
* Are at least 13 years old (need consent if under 18).
* Are in reasonably good health.
* Are expected to live for at least 6 months.
* Are receiving anti-HIV medications at study entry.

Exclusion Criteria

You will not be eligible for this study if you:

* Have/had MAC disease.
* Have been unable to take azithromycin in the past.
* Are on any medications that act against MAC.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 850
Dates: Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa El-Sadr, Study Chair; William Burman, Study Chair
Locations (19):
- United States (19):
  - Community Consortium / Jon Kaiser Wellness Ctr, San Francisco, California
  - Community Consortium / UCSF, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Washington Reg AIDS Prog / Dept of Infect Dis, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - LSMUC / Lions Clinic, New Orleans, Louisiana
  - Catherine McAuley Health Ctr, Detroit, Michigan
  - Wayne State Univ - WSU/DMC / Univ Hlth Ctr, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Cln Trials / Dept of Med, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners in Research / New Mexico, Albuquerque, New Mexico
  - Harlem AIDS Treatment Grp / Harlem Hosp Ctr, New York, New York
  - The Research and Education Group, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Saint Joseph's Hosp, Philadelphia, Pennsylvania
  - Richmond AIDS Consortium / Div of Infect Diseases, Richmond, Virginia

REFERENCES:
- [Background] Burman W, El-Sadr W, Grant L, Matts J, Zeh D, Gallagher B, Hafner R, Crane L, Gordin F. Low rates of all opportunistic infections among patients with advanced HIV disease responding to antiretroviral therapy - the CPCRA 048 Cohort. 7th Conf Retroviruses Opportunistic Infect. 2000 Jan 30-Feb 2 (abstract no 241)
- [Background] El-Sadr WM, Manneheimer S, Grant L, Matts J. Use of PCP and MAC prophylaxis among eligible patients with and without CD4+ rebound. 39th Intersci Conf Antimicrob Agents Chemother. 1999 Sept 26-29
- [Background] El-Sadr WM, Burman W, Grant L, Matts JP, Zeh D, Crane L, Gallagher B, Gordin F, Hafner R. Prophylaxis for Mycobacterium avium Complex can be deferred among patients with a past CD4 count <50 cells/mm3 who responded to antiretroviral therapy: results of a placebo-controlled trial (CPCRA 048). 7th Conf Retroviruses Opportunistic Infect. 2000 Jan 30-Feb 2 (abstract no 247)
- [Background] El-Sadr WM, Burman WJ, Grant LB, Matts JP, Hafner R, Crane L, Zeh D, Gallagher B, Mannheimer SB, Martinez A, Gordin F. Discontinuation of prophylaxis against Mycobacterium avium complex disease in HIV-infected patients who have a response to antiretroviral therapy. Terry Beirn Community Programs for Clinical Research on AIDS. N Engl J Med. 2000 Apr 13;342(15):1085-92. doi: 10.1056/NEJM200004133421503. PMID 10766581